CLINICAL TRIAL: NCT00780195
Title: Metabolic Adaptations to Diabetes
Brief Title: Metabolic Adaptations to Diabetes in African Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Steve Davis, Department Chair, Vanderbilt University
Allocation: Randomized | Model: Factorial | Masking: Single
Other Study IDs: IRB # 8177
Record Dates: First submitted 2008-10-24; First posted 2008-10-27 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Diabetes
Keywords: hypoglycemia; African Americans
MeSH Terms: conditions — Diabetes Mellitus; Hypoglycemia | interventions — Glucose Clamp Technique

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Single 2 hour hyperinsulinemic euglycemic clamp study at ~90 mg/dl.
  Interventions: Procedure: glucose clamp
- 2 (Experimental): Single 2 hour hyperinsulinemic hypoglycemic clamp study at ~70 mg/dl.
  Interventions: Procedure: glucose clamp
- 3 (Experimental): Single 2 hour hyperinsulinemic hypoglycemic clamp at ~60 mg/dl.
  Interventions: Procedure: glucose clamp
- 4 (Experimental): Single, 2 hour hyperinsulinemic hypoglycemic clamp at ~50 mg/dl.
  Interventions: Procedure: glucose clamp

INTERVENTIONS:
Procedure: glucose clamp — 2 hour hyperinsulinemic euglycemic clamp (90 mg/dl)
  Arms: 1
Procedure: glucose clamp — 2 hour hyperinsulinemic hypoglycemic clamp (70 mg/dl)
  Arms: 2
Procedure: glucose clamp — 2 hour hyperinsulinemic hypoglycemic clamp (60 mg/dl)
  Arms: 3
Procedure: glucose clamp — 2 hour hyperinsulinemic hypoglycemic clamp (50 mg/dl)
  Arms: 4

SUMMARY:
We do not know why diabetic patients cannot protect themselves against low blood sugar. Therefore, in this study, we will perform a comprehensive assessment of the body's response to low blood sugar by measuring changes in blood hormones, blood sugar production, and nerve signals.

DETAILED DESCRIPTION:
Morning and afternoon hypoglycemic episodes of 70, 60, or 50 mg/dl produce increased blunting of subsequent counterregulation dependent upon the depth of preceding hypoglycemia. We wanted to test this hypothesis in healthy African American individuals to determine if there is a difference in their responses to varying depths of hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females aged 18-40 yrs with no family history of diabetes mellitus.
* All prospective volunteers will have routine blood tests to screen for biochemical, hormonal and hematological abnormalities.
* Female volunteers will also undergo an HCG urine pregnancy test.

Exclusion Criteria:

* Prior or current history of poor health
* Abnormal results following blood and physical examination
* Pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 1998-07; Primary Completion 2000-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
catecholamines | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Stephen N. Davis, MD, Principal Investigator — Vanderbilt University